CLINICAL TRIAL: NCT06174168
Title: Combining Modified Frailty Index 11 (MFI-11) in Predicting Complements in Patients Over 65 Years of Age Who Underwent Endobronchial Ultrasonography-guided Transbronchial Needle Aspiration (EBUS-TBNA) Under Sedation.
Brief Title: The Decisiveness of MFI-11 in Predicting Complications in Patients > 65 Years Who Underwent EBUS-TBNA Under Sedation
Status: Completed | Type: Observational
Sponsor: Ankara Ataturk Sanatorium Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Irem Ulutas Ordu, RESEARCHER MD, Ankara Ataturk Sanatorium Training and Research Hospital
Other Study IDs: E-53610172-799-224037416
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Sedation Complication; EBUS Guided Transbronchial Needle Aspiration; Monitored Anesthesia Care; Elderly Patients
Keywords: sedation; ebus guided transbronchial needle aspiration; monitored anesthesia care; elderly patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Patients who did not develop any complication in the EBUS-TBNA. Patients may experience intraoperative complications (bleeding, hypoxemia, hypotension, arrhythmia, bronchospasm, pneumothorax, subcutaneous emphysema/mediastinal emphysema, respiratory depression), and postoperative complications (bleeding, pneumonia, respiratory failure, atelectasis, pleural effusion/empyema, pulmonary embolism, pulmonary edema). Complications that develop (such as acute respiratory distress syndrome, delirium, and mortality) will be recorded. After the procedure, any complications that may develop in the patients within 30 days will be questioned and recorded.
  Interventions: Other: Modified Frailty Index -11
- Group 2: Patients who developed complications during EBUS-TBNA. Patients may experience intraoperative complications (bleeding, hypoxemia, hypotension, arrhythmia, bronchospasm, pneumothorax, subcutaneous emphysema/mediastinal emphysema, respiratory depression), and postoperative complications (bleeding, pneumonia, respiratory failure, atelectasis, pleural effusion/empyema, pulmonary embolism, pulmonary edema). Complications that develop (such as acute respiratory distress syndrome, delirium, and mortality) will be recorded. After the procedure, any complications that may develop in the patients within 30 days will be questioned and recorded.
  Interventions: Other: Modified Frailty Index -11

INTERVENTIONS:
Other: Modified Frailty Index -11 — MFI-11: the parameter included in the score is history of congestive heart failure, presence of diabetes mellitus, history of chronic obstructive pulmonary disease or pneumonia, functional health status/dependence, history of hypertension, history of myocardial infarction, cardiac problems, cognitive impairment, history of transient ischemic attack or cerebrovascular accident, history of peripheral vascular disease is questioned. Patients will be monitored according to standard non-operating room anesthesia procedures.
  Other Names: MFI-11

SUMMARY:
The aim is to evaluate the feasibility of MFI-11, one of the comprehensive frailty tests, before EBUS-TBNA. The secondary aim is to evaluate the usefulness of MFI-11 in predicting complications in risk assessment before EBUS-TBNA.

DETAILED DESCRIPTION:
Patients who will receive anesthesia are directed to the anesthesia clinic for preoperative evaluation. The primary purpose of preoperative assessment is to reduce perioperative morbidity and increase quality, reduce the cost of perioperative care, and ensure that the patient recovers as quickly as possible. In this context, the American Society of Anesthesiology (ASA) score is a classification that includes medical comorbidities. The classification system alone does not predict perioperative risks, but when combined with other factors (e.g. type of surgery, frailty) it may help predict perioperative risks. Age is not among the criteria in the ASA.

In elderly patients, the indicator of decreased reserves and resulting weakness is called "frailty". Frailty is considered vulnerability and functional impairment caused by a significant decline in multiple systems. Objective, repeatable, and accepted scales must be used when evaluating frailty. MFI-11 is a strong predictor of mortality and postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent EBUS-TBNA under sedation
* Patients aged >65 years
* ASA 1-3 patients

Exclusion Criteria:

* Patients who did not volunteer for the study
* < 65 years old patients
* ASA > 3 patients
* Patients with psychiatric illness
* Intubated patients
* Patients with tracheostomy
* Patients with body mass index > 30 kg/m2
* Patients with nasal and nasopharyngeal disease
* Patients with drug allergies (drugs used in anesthesia)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: EBUS-TBNA planned >65 years of age, including ASA 1-3 parts. The estimated duration is expected to be three months. Patients with a body mass index over 30 kg/m2, intubation or tracheostomy, nasal or nasopharyngeal disease, communication difficulties, ASA 4-5 patients, psychiatric illnesses, and emergency diseases will be excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Modified Fraility Index -11 | Preoperative 1 time
  In elderly patients, the indicator of decreased reserves and resulting weakness is called "frailty". Frailty is considered vulnerability and functional impairment caused by a significant decline in multiple systems. When evaluating frailty, objective, repeatable and accepted scales must be used. MFI-11 is a strong predictor of mortality and postoperative complications. MFI-11 is calculated by dividing the existing deficits by the total number of deficits. Each parameter is 1 point, and the MFI-11 score will be calculated by adding all the points and dividing by 11. The higher this score, the more frail the patient. As a result of studies comparing frailty, if the MFI-11 score is greater than ≥ 0.27, these patients are defined as frail.

CONTACTS AND LOCATIONS:
Overall Officials: İrem ULUTAŞ ORDU, M.D, Principal Investigator — Ankara Atatürk Sanatoryum Training and Research Hospital
Locations (1):
- Ankara Atatürk Sanatoryum Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No